CLINICAL TRIAL: NCT01317095
Title: A Prospective Randomized Study of Two Types of Sternal Closure After Open Heart Surgery: Rigid Sternal Fixation vs. Sternal Wire Closure
Brief Title: A Study of Sternal Closure After Open Heart Surgery: Rigid Versus Wire Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sternal Closure
Record Dates: First submitted 2011-03-10; First posted 2011-03-17 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-01

CONDITIONS: Pain
Keywords: Rigid fixation; Sternal closure; Open heart surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Wire closure is the intervention (Active Comparator): Patients will have their sternum closed using stainless steel wires.
  Interventions: Device: Sternalock Rigid Fixation
- Rigid fixation (Active Comparator): Patients will have their sternum closed by rigid fixation using Starnalock plates.
  Interventions: Device: Sternalock Rigid Fixation

INTERVENTIONS:
Device: Sternalock Rigid Fixation — Patients will have their sternum closed by rigid fixation using Sternalock plates.

SUMMARY:
The investigators are conducting this research to compare two different methods of closure of the sternum after cardiac surgery to determine if one method is better than the other. Open heart surgery always requires a sternotomy, and at the end of surgery the sternum needs to be closed. The sternum can be closed with Stainless Steel Wires or Sternalock rigid sternal closure system with equivocal results; however, the outcomes of these two methods have never been investigated in a randomized study. Thus, the investigators are conducting this study to compare two different methods of closure if one method demonstrates any recovery benefit over the other, using randomizing the subjects 1:1 to either rigid fixation with Sternalock or stainless steel wire closure. Recover benefit will be measured by postoperative intubation time, length of intensive care unit stay, and overall postoperative length of stay

DETAILED DESCRIPTION:
1. Subjects:

   Inclusion criteria:
   1. scheduled (elective or urgent) coronary artery bypass graft with or without valvular surgery by our cardiothoracic surgery division.
   2. patient age ≥18 and <80 .
   3. patient undergoing elective surgery.
   4. patient undergoing urgent surgery (defined as surgery scheduled while the patient is in the hospital and performed during the same hospital admission with stable medical condition)
   5. patients who is willing to sign the informed consent to participate the study.

   Pre- operative exclusion criteria:
   1. patient undergoing redo-sternotomy.
   2. patient undergoing emergent surgery (defined as life-threatening or unstable condition requiring surgery on the same day of the surgical consultation.)
   3. patients on dialysis
   4. patients undergoing ventricular assist device insertion, transplant surgery, or aortic surgery.
   5. patients with body mass index ≥ 40.
   6. patients with active endocarditis.
   7. patients with known metal allergy.
   8. patient who refuses consent.
   9. patient who is unable to follow the postoperative instructions.

   Intraoperative exclusion criteria:
   1. osteoporosis or poor quality of sternum.
   2. unstable sternal fracture.
   3. sternum too thin (less than 4 mm) or too thick (greater than 14 mm) as determined by direct measurement.
   4. bilateral mammary artery harvest (causing poor blood supply to the sternum).
   5. patients in whom the chest needs to be left open due to medical reasons.
2. Procedures:

   Preoperative testing, medical evaluation, cardiac surgery and postoperative care will all be performed per standard of care. The patients will sign a separate consent for their open heart surgery.

   Baseline screening: Medical history and preoperative testing are reviewed to determine if the patient is a suitable candidate of the study. If the patient meets inclusion criteria, the study will be explained and the two closure methods will be discussed; it will be explained that the method of sternal closure will be determined by randomization if they choose to participate in the study. If they still want to participate, the consent will be signed.

   Randomization procedure: On the day of heart surgery, subjects will be randomized 1:1 to either closure with stainless steel wires or rigid closure with Sternalock System by opening an envelope in the operating room. After randomization, if the patient meets any of the intraoperative exclusion criteria the patient will be excluded from the study.

   Data collection: Ventilator time, length of intensive care unit stay and length of hospital stay will be collected. Daily 6 am pain VAS (visual analog scores) scores will be collected while the patient is hospitalized. Complications such as sternal infection, sternal dehiscence, pneumonia will be monitored.

   Follow-up visit: At a routine postoperative follow-up visit, usually occurring at 4-8 weeks after surgery, sternal stability and pain scores will be assessed.
3. Data analysis:

Plan is 2 group comparisons using student t-tests or chi-square tests performed to identify the factors contributing to intubation time, ICU stay and hospital stay. Univariate analysis followed by multivariate analyses to identify independent risk factor will be performed by statistical package (JMP software)

ELIGIBILITY:
Inclusion Criteria:

1. scheduled (elective or urgent) coronary artery bypass graft with or without valvular surgery by our cardiothoracic surgery division.
2. patient age ≥18 and <80 .
3. patient undergoing elective surgery.
4. patient undergoing urgent surgery (defined as surgery scheduled while the patient is in the hospital and performed during the same hospital admission with stable medical condition)
5. patients who is willing to sign the informed consent to participate the study.

Exclusion Criteria:

Pre- operative exclusion criteria:

1. patient undergoing redo-sternotomy.
2. patient undergoing emergent surgery (defined as life-threatening or unstable condition requiring surgery on the same day of the surgical consultation.)
3. patients on dialysis
4. patients undergoing ventricular assist device insertion, transplant surgery, or aortic surgery.
5. patients with body mass index ≥ 40.
6. patients with active endocarditis.
7. patients with known metal allergy.
8. patient who refuses consent.
9. patient who is unable to follow the postoperative instructions.

Intraoperative exclusion criteria:

1. osteoporosis or poor quality of sternum.
2. unstable sternal fracture.
3. sternum too thin (less than 4 mm) or too thick (greater than 14 mm) as determined by direct measurement.
4. bilateral mammary artery harvest (causing poor blood supply to the sternum).
5. patients in whom the chest needs to be left open due to medical reasons.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-03; Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hitoshi Hirose, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Division of Cardiothoracic Surgery, Thomas Jefferson University — http://hospitals.jefferson.edu/departments-and-services/cardiothoracic-surgery.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rigid Fixation | Wire Closure is the Intervention
Started | 39 | 41
Completed | 39 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wire Closure is the Intervention | Rigid Fixation | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 19 | 34
  >=65 years | 26 | 20 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (9) | 65 (8) | 65 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 34 | 31 | 65
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 39 | 80

OUTCOME MEASURES:

1. Primary Outcome: Intubation Time
Description: The primary objective of this study is to determine if rigid sternal fixation can shorten the postoperative intubation time after open heart surgery compared to the wire closure
Time Frame: 48 hours after surgery
Population: Intubation time
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Wire Closure: Patients will have their sternum closed using stainless steel wires.
Arm/Group | Rigid Fixation | Wire Closure
Number analyzed (Participants) | 39 | 41
hours | 7 (5) | 9 (9)

2. Secondary Outcome: Pain Scores.
Description: One of the secondary outcomes are monitoring the patient's pain scores from postoperative day 1 till day 5.
Time Frame: 5 days after surgery
Population: Likert Pain Scale from 0-10 (0: no pain; 10:worst possible pain)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rigid Fixation | Wire Closure
Number analyzed (Participants) | 39 | 41
score on a scale
  Pain score on day1 | 2.3 (3.1) | 2.8 (3.4)
  Pain score on day2 | 2.2 (2.7) | 2.0 (2.7)
  Pain score on day3 | 0.5 (1.4) | 0.8 (1.7)
  Pain score on day4 | 0.5 (1.8) | 1.7 (3.4)
  Pain score on day5 | 0.2 (1.0) | 0.4 (1.3)

3. Secondary Outcome: Length of ICU Stay
Description: Length of postoperative intensive care unit stay.
Time Frame: ICU stay
Population: Postoperative average intensive care unit stay (hours)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Rigid Fixation | Wire Closure
Number analyzed (Participants) | 39 | 41
hours | 51 (29) | 55 (44)

4. Secondary Outcome: Postop Length of Hospital Stay.
Description: Postoperative length of hospital stay.
Time Frame: Until hospital discharge
Population: Postoperative length of hospital stay.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Rigid Fixation | Wire Closure
Number analyzed (Participants) | 39 | 41
days | 7 (4) | 8 (7)

ADVERSE EVENTS:
Arm/Group | Wire Closure is the Intervention | Rigid Fixation
All-Cause Mortality (participants affected / at risk) | 1/41 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/41 | 1/39
Other Adverse Events (participants affected / at risk) | 0/41 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wire Closure is the Intervention (N=41) | Rigid Fixation (N=39)
Deep sternal infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — One patient developed deep sternal infection. Patient was treated with antibiotics and muscle flap, then eventually discharged from hospital
Mortality (Nervous system disorders) | 1 (1) | 0 (0) — Mortality due to acute stroke

LIMITATIONS AND CAVEATS:
Small number of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes